CLINICAL TRIAL: NCT07390812
Title: Respiratory Transition Without Continuous Positive Airway Pressure in Term Infants With Mild Respiratory Distress: A Pilot Study
Brief Title: Respiratory Transition Without Continuous Positive Airway Pressure
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2022-0654
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Mild Respiratory Distress
Keywords: mild respiratory distress; term neonates; continuous positive airway pressure
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Continuous positive airway pressure (CPAP) is administered for mild respiratory distress
  Interventions: Other: CPAP
- Watchful waiting (Experimental): Neonates with mild respiratory distress are observed for 20 minutes, and CPAP is administered at 25 minutes of life if respiratory distress continues or earlier if moderate to severe respiratory distress occurs
  Interventions: Other: Transition without Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Other: Transition without Continuous Positive Airway Pressure (CPAP) — Allowing transition without CPAP administration was assessed at 25 minutes of life
  Arms: Watchful waiting
Other: CPAP — CPAP administration as per standard of care
  Arms: Standard of care

SUMMARY:
The primary aim of this research project is to determine if term neonates (37:0 to 41:6 weeks' gestational age) with mild respiratory distress can safely transition without continuous positive airway pressure (CPAP). The secondary aim is to determine the incidence of pneumothorax (PTX) for all term neonates assessed to have mild respiratory distress in the delivery room (DR).

ELIGIBILITY:
Inclusion Criteria:

* Full term infants (37 weeks + 0days to 41 weeks +6days gestational age)
* Born via scheduled c-sections without labor
* Who develop mild respiratory distress, defined as nasal flaring or, intermittent grunting, and/or mild retractions and/or +/- mild tachypnea ( respiratory rate 61-90).

Exclusion Criteria:

* Moderate to severe respiratory distress (continuous grunting, or moderate retractions or respiratory rate greater than 90 breaths per minute),
* need for positive pressure ventilation (PPV) or advanced resuscitation in the first 5 minutes of life,
* meconium stained amniotic fluid,
* major congenital anomalies or chromosomal abnormalities.

Ages: 37 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Need for CPAP use at 25 minutes of life | At 25 minutes post birth (after 20 minutes of observation)
  Babies with mild respiratory distress will be observed for 20 minutes (randomized at 5 minutes of life) using a pulse oximeter (per institutional post-resuscitation care guidelines) and under the study team's direct observation.
  The active cohort will not receive CPAP unless respiratory distress worsens.

SECONDARY OUTCOMES:
Prevalence of pneumothorax in neonates | Within 6 hours of life
  Number of babies with pneumothorax in neonates as assessed by a chest ultrasound.
NICU (Neonatal Intensive Care Unit) admission during hospital stay | Hospital day (from birth to discharge)
  Number of babies admitted to the NICU for respiratory distress during the initial hospital stay (on average, 1-4 days).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Spillane, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univeristy Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No